CLINICAL TRIAL: NCT03256279
Title: Comparison of Mechanical Properties and Clinical Efficacy Between Heat-activated and Superelastic Nickel-Titanium (NiTi) Archwires.
Brief Title: Mechanical Properties and Clinical Efficacy of Two Nickel-Titanium (NiTi) Archwires
Acronym: (NiTi)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Universitaria CIEO (Other)
Responsible Party: Principal Investigator, Suly Amaya, Teacher Orthodontic department, Fundación Universitaria CIEO
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UniCIEO
Record Dates: First submitted 2017-08-16; First posted 2017-08-22 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Crowding of Anterior Mandibular Teeth
Keywords: Orthodontic Wires; Alloys/therapeutic use; Orthodontics, corrective

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Only one of the investigators are going to know the archwire assigment, the other ones who are going to do the measures are going to be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat-activated archwire (Experimental): .014" NiTi heat-activated archwire in the lower arch during the first three months of the orthodonci treatment
  Interventions: Device: .014" NiTi heat-activated archwire
- superelasticwire (Active Comparator): This arm are going to receive .014" NiTi Superelastic archwire in the lower arch during the first three months of the orthodonci treatment
  Interventions: Device: .014" NiTi Superelastic archwire

INTERVENTIONS:
Device: .014" NiTi heat-activated archwire — .014" NiTi heat-activated archwire In the lower arch during the first three months of the orthodonci treatment
  Arms: Heat-activated archwire
Device: .014" NiTi Superelastic archwire — .014" NiTi superelastic archwireIn the lower arch during the first three months of the orthodonci treatment
  Arms: superelasticwire

SUMMARY:
Objective: to compare the changes of the mechanical properties measured by tensile test and three point bending test of two NiTi archwires (heat-activated and superelastic); when exposed to the oral conditions during the first three months of orthodontic treatment and to evaluated their clinical efficacy in lower arch crowding resolution in the anterior mandibular arch.

Methods: Randomized clinical trial in 54 orthodontic patients with moderate crowding. They are going to be randomly assigned in to two intervention groups, each group with 27 patients. One group are going to be treated with heat-activated NiTi archwires and the other group with superelastic NiTi archwires. The patients are going to be followed up for three months and cast models will be taken every month. Measures of anterior lower arch crowding resolution are going to be taken by previously-calibrated operators. Six archwires of each group will be chosen at random and will have tensile test and three-point bending test and the mechanical properties are going to measure before and after its clinical use. The outcomes are going to be determined and compared between groups, with correspondent statistical test and the results are going to be analyzed.

DETAILED DESCRIPTION:
PICO QUESTION:

* Does the amount of the resolution of the anterior lower arch crowding increase in the patients with superelastic NiTi archwire compared with the patients with heat-activated NiTi archwire during the first three months of orthodontic treatment and/or its mechanical properties change after three months of clinical use?

Population: Orthodontic patients with moderate anterior mandibular crowding Intervention: .014" Superelastic NiTI archwire (3M Unitek, Monrovia, CA) Comparison: .014" Heat activated NiTi archwire (3M Unitek, Monrovia, CA)

Outcomes:

Primary Outcomes:

* Quantity of resolution of anterior mandibular crowding every month for three months
* Mechanical properties measured by tensile test and three point bending test before and after the three first months of orthodontic treatment.

Secondary Outcomes: Archwires deformation under oral conditions during the first three months of the orthodontic treatment.

AIMS

GENERAL AIM To compare the changes of the mechanical properties measured by tensile test and three point bending test of two NiTi archwires (heat-activated and super-elastic); when exposed to the oral conditions during the first three months of orthodontic treatment and to evaluated the clinical efficacy in lower anterior arch crowding resolution.

SPECIFIC AIMS

* To recruit 54 orthodontic patients, 13-25 years old, without extraction into a randomized clinical trial design, single-blinded trial, into the effects of NiTi arch-wires alloy in the resolution of the anterior mandibular crowding during the three first months of the orthodontic treatment.
* To test the hypothesis that, compared the resolution of the anterior mandibular crowding in the first three months of orthodontic treatment, with those to receive NiTi heat-activated arch-wire, those assigned to receive superelastic NiTi archwire
* More amount of resolution of the anterior mandibular crowding
* Differences in the changes of mechanical properties after clinical use
* Less archwire deformation

METHODS

OVERVIEW OF DESIGN Study Design: Randomized clinical trial

* Randomized clinical trial in 54 orthodontic patients with moderate crowding. They are going to be randomly assigned in to two intervention groups, each group with 27 patients. One group are going to be treated with heat-activated NiTi archwires and the other group with super-elastic NiTi archwires.
* Blinding: It is not possible to blind patients and clinical staff, but we are going to blind the operators who will perform the measurements and the data analysis (single-blinded).

We are going to have an exact clinical protocol for both groups with the only difference being in the NiTI arch-wire alloy.

MBT prescription .022 slot. Alginate impressions and cast models at the beginning of the study, immediately after the first, second and third month of the orthodontic treatment.

Measures of anterior lower arch crowding resolution are going to be taken by previously-calibrated operators.

Arch-wires deformation are going to be evaluated by visual observation every month in monthly clinical visits.

The measures of the mechanical properties measured by tensile test and three point bending test of two NiTi archwires (heat-activated and super-elastic); are going to take before and after the first three months of orthodontic treatment.

DESIGN FOR SAMPLING

Study Population:

- Orthodontic patients from the orthodontic department clinic of the UniCIEO

Sampling:

* No probabilistic: convenience sample
* Consecutive sample of consenting patients

PLANS FOR RECRUITMENT

Patients of the Clinic University (UniCIEO) that meet the selection criteria and accept to participate.

MEASUREMENTS

MAIN PREDICTOR VARIABLE

- Type of NiTi Alloy used (NiTi superelastic arch-wire; NiTi heat-activated arch-wire)

POTENCIAL CONFOUNDING VARIABLES - Age

- Sex

OUTCOME VARIABLES

Plaster models Outcomes:

- Quantity of anterior mandibular crowding resolution measured monthly

Mechanical Properties Outcomes:

- Measured in vitro with an Instrom before and after three months of the orthodontic treatment by tensile test and three point bending test

Archwire Outcomes:

- Archwire deformation measure at monthly visit, by visual evaluation

STATISTICAL ISSUES

APPROACH TO STATISTICAL ANALYSIS

The data will be processed in the statistics program Stata 14 (Stata Corp 2011. Stata Statistical Software: Release 14. College Station, TX: Stata Corp LP). Qualitative variables are going to be described by frequencies and percentages; quantitative variables will resume as average and standard deviation. The association between qualitative variables will be calculated by Chi-square test. For two group comparisons, we are going to use the t test or Wilcoxon-Mann-Whitney test. Significance level is going to be set at P<0.05.

HYPOTHESIS, SAMPLE SIZE AND POWER

Hypothesis:

Null Hypothesis H0: compared the resolution of the anterior mandibular crowding in the first three months of orthodontic treatment, with those to receive NiTi heat-activated archwire, those assigned to receive superelastic NiTi archwire

* Same amount of resolution of the anterior mandibular crowding
* Same changes in mechanical properties after clinical use
* Same archwire deformation

Alternate Hypothesis Ha: compared the resolution of the anterior mandibular crowding in the first three months of orthodontic treatment, with those to receive NiTi heat-activated archwire, those assigned to receive superelastic NiTi archwire

* More amount of resolution of the anterior mandibular crowding
* Differences in the changes of mechanical properties after clinical use
* Less archwire deformation

Sample size calculation and power:

It was calculated with the software Epidat (software Epidat version 4.1). With 90% power and a 5% level of significance and with standard deviation data from a previous study, the sample should comprise at least 27 patients per group.

QUALITY CONTROL AND DATA MANAGEMENT

Bias Control:

Selection bias:

- Randomization

Information bias:

* The principal investigators are going to train the observers in the theoretical and practical issues of all the measures of the variables of this study developing an operations manual.
* The observers are going to be calibrated and evaluated in intra and extra observer concordance by Bland Altman plot with previously fixed acceptable limits.
* All variables, are going to be re-measured after two weeks in subjects randomly selected.
* Random and systematic errors are going to be calculated with Dahlberg´s formula and dependent t test, respectively.
* Same clinical protocol for groups, the only difference in the intervention. All clinical and laboratory procedures will meet quality standards. The research team will take care of the data in order to be reliable and accurate The research team will take care that complete and accurate records will be maintained Statistical methods are going to be pre-specified and carefully followed The results are going to be clearly and fairly reported

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic treatment without extraction with moderate anterior mandibular crowding (little index: 4-6mm)
* Age range between 15-25 years' old
* Non gingivitis or untreated caries at the start of orthodontic treatment
* Not need for intermaxillary elastics, striping, open compressed Nit springs, active labial arch, stainless ligature, during the first to the third months of orthodontic treatment
* Complete orthodontic appliances in the lower arch (at minimum from first molar to the first molar)

Exclusion criteria:

* Patients with systemic disease
* Medicated patients (long term use of antibiotics, Phenytoin, cyclosporine, anti- inflammatory drugs, systemic corticosteroids, and calcium channel blockers)
* Diseases that may affect dental movement
* Syndromic patients
* Patients with a history of trauma and/or root resorption at the lower arch
* Patients who do not attend more than one month to the appointment
* Lower .014" NiTi archwires that fracture during the first three months of the study.
* Patients with previous orthodontic treatment

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2017-07-08 (Actual); Primary Completion 2019-12-10 (Estimated); Study Completion 2019-12-10 (Estimated)

PRIMARY OUTCOMES:
Quantity of anterior mandibular crowding resolution | baseline and three months
  MBT prescription .022 slot. Alginate impressions and cast models at the beginning of the study, immediately after the first, second and third month of the orthodontic treatment.
  Measures of anterior lower arch crowding resolution are going to be taken by previously-calibrated operators.

SECONDARY OUTCOMES:
Changes in Mechanical properties | baseline and three months
  Mechanical properties of six archers random choose per group are going to be measured by tensile test and three-point bending test, before and three months after clinical use.
Archwire deformation | baseline and three months
  Archwire deformation will be measure by visual evaluation, each month of clinical use

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Plaza, Ms., Study Director — Fundación Universitaria CIEO
Locations (1):
- Orthodontic clinic of Post-graduation program UniCIEO, Bogotá, Bogotá D. C., Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amaya Gonzalez SY, Roncancio AP, Acuna EA, Guevara Barreto LA, Vargas NM, Plaza-Ruiz SP. Alignment efficiency of heat activated and superelastic nickel-titanium archwires in orthodontic patients over three months: A Single-center, randomized clinical trial. J Orthod Sci. 2023 Mar 18;12:9. doi: 10.4103/jos.jos_19_22. eCollection 2023. PMID 37351408